CLINICAL TRIAL: NCT06406829
Title: Perioperative Multimodal Analgesia Protocol for Supratentorial Craniotomy：a 2× 2 Factorial Randomized Clinical Trial
Brief Title: Perioperative Multimodal Analgesia Protocol for Supratentorial Craniotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Deputy chief of Department of Anesthesiology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024007
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pain; Analgesia; Supratentorial Brain Tumor
Keywords: multimodal analgesia; Postoperative acute pain
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Local analgesic techniques + dexmedetomidine group (Experimental): The patients in this group will be received scalp nerve block before surgery with 0.67 % liposomal bupivacaine. The patients also will be given dexmedetomidine intravenously at a rate of 0.4 μg/kg/h from skin incision until the beginning of dura mater closure, and will be adjusted to 0.05 μg/kg/h for 48 hours after surgery.
  Interventions: Drug: Dexmedetomidine; Other: Local analgesic techniques
- Local analgesic techniques and placebo dexmedetomidine group (Experimental): The patients in this group will be received scalp nerve block before surgery with 0.67 % liposomal bupivacaine. For dexmedetomidine placebo group, normal saline will be infused at the same rate as dexmedetomidine during surgery and for 48 hours after surgery.
  Interventions: Drug: Normal saline; Other: Local analgesic techniques
- Placebo local analgesic techniques and dexmedetomidine group (Experimental): The patients in this group will not receive scalp nerve block. The patients will be given dexmedetomidine intravenously at a rate of 0.4 μg/kg/h from skin incision until the beginning of dura mater closure, and will be adjusted to 0.05 μg/kg/h for 48 hours after surgery.
  Interventions: Drug: Dexmedetomidine; Other: no Local analgesic techniques
- Placebo local analgesic techniques and placebo dexmedetomidine group (Placebo Comparator): The patients in this group will not receive scalp nerve block before surgery . For dexmedetomidine placebo group, normal saline will be infused at the same rate as dexmedetomidine group during surgery and for 48 hours after surgery.
  Interventions: Drug: Normal saline; Other: no Local analgesic techniques

INTERVENTIONS:
Drug: Dexmedetomidine — The 200ug dexmedetomidine will be diluted into a 50ml syringe and administered with 0.4ug/kg/h intraoperatively and 0.05 μg/kg/h for 48 hours after surgery.
  Other Names: DEX
  Arms: Local analgesic techniques + dexmedetomidine group; Placebo local analgesic techniques and dexmedetomidine group
Drug: Normal saline — In the placebo group, the 0.9% saline is administered with the same volume at the same speed as the dexmedetomidine group
  Other Names: NS
  Arms: Local analgesic techniques and placebo dexmedetomidine group; Placebo local analgesic techniques and placebo dexmedetomidine group
Other: Local analgesic techniques — As for scalp nerve block, each nerve will be blocked separately with 1-2 mL of 0.67 % liposomal bupivacaine
  Other Names: LAT
  Arms: Local analgesic techniques + dexmedetomidine group; Local analgesic techniques and placebo dexmedetomidine group
Other: no Local analgesic techniques — No Local analgesic techniques will be given.
  Other Names: NLAT
  Arms: Placebo local analgesic techniques and dexmedetomidine group; Placebo local analgesic techniques and placebo dexmedetomidine group

SUMMARY:
Supratentorial craniotomy is one of the most common neurosurgical procedures, with severe perioperative pain. Inadequate perioperative pain relief has been associated with increased blood pressure and intracranial pressure, favoring bleeding and cerebral cerebral hypoperfusion. The ideal analgesia for neurosurgery requires complete pain relief, eliminates the side effects of opioid drugs and no influence for neurological function. Previous studies have proposed a multimodal analgesic strategy, combining analgesics and local anaesthesia, it is expected to achieve the above benefits.

DETAILED DESCRIPTION:
The trial has been designed to analyze the efficacy of local analgesic techniques and dexmedetomidine in the treatment of postoperative acute pain in craniotomy. This randomized clinical trial aims to enroll 2000 patients, which will be randomized to one of 4 groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 65 years
* American Society of Anesthesiologists physical status I to III
* Scheduled to undergo elective supratentorial tumor resection

Exclusion Criteria:

* Incision-area skin infection
* A history of previous craniotomy
* Allergy to study medications
* A history of preoperative change in consciousness or cognitive function
* Severe hepatic or renal dysfunction
* Severe bradycardia (heart rate<40 beats/min)
* Sick sinus syndrome or second- to-third degree atrioventricular block

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative amount of sufentanil used by patient-controlled analgesia (PCIA) in patients within 48 hours postoperatively. | 48 hours postoperatively
  Cumulative amount of sufentanil used by patient-controlled analgesia (PCIA) in patients within 48 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Peng, Dr, Principal Investigator — Beijing Tiantan Hospital